CLINICAL TRIAL: NCT02234713
Title: Treatment Adherence in Pediatric Multiple Sclerosis
Brief Title: Adherence in Pediatric Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: National Multiple Sclerosis Society (Other); Loma Linda University (Other); University of Pittsburgh (Other); Children's Hospital of Philadelphia (Other); Boston Children's Hospital (Other); Baylor College of Medicine (Other); University of Alabama at Birmingham (Other); Mayo Clinic (Other); University of Colorado, Denver (Other); University of California, San Francisco (Other); Washington University School of Medicine (Other); Alberta Children's Hospital (Other); The Cleveland Clinic (Other); DeltaQuest Foundation (Unknown)
Responsible Party: Principal Investigator, E. Ann Yeh, Staff Neurologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1000035924; HC 0148 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Behavioural Intervention/Feedback (Experimental): The behavioral interventionist will contact the patient and parent by email and telephone to schedule a telephone call to review the downloaded adherence information and discuss barriers experienced by the patient/parent using a standard script. The behavioral feedback will be administered three times: at 1-, 2- and 3-months post-baseline.
  Interventions: Behavioral: Motivational Interview
- Video Attention Control (Active Comparator): The patients in this arm of the study will be emailed a link to an educational video about Pediatric MS and therapy for MS at three time points: 1-, 2-, and 3-months post-baseline.
  Interventions: Other: Video Attention Control

INTERVENTIONS:
Behavioral: Motivational Interview
  Arms: Behavioural Intervention/Feedback
Other: Video Attention Control
  Arms: Video Attention Control

SUMMARY:
Disease modifying therapies (DMT) are widely used for children and adolescents with MS. Nonetheless, many pediatric patients continue to relapse and therefore require changes in therapy. We designed this research study to learn more about medication use in children and adolescents with MS. We are also interested in learning what a behavioral feedback intervention can tell us about adherence to medicine. Finally, we hope this research project will inform the way we provide clinical care for children and adolescents with MS.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent boys/girls who are 10 to 17 years 11 months old;
* Have a diagnosis of MS, as per revised McDonald diagnostic criteria and International Pediatric MS Study Group criteria;
* Prescribed with an oral or injectable disease-modifying therapy for MS for at least six months.

Exclusion Criteria:

* Have non-specific white matter abnormalities and metabolic or infectious etiologies for white matter abnormalities. This is indicative of not having a true diagnosis of MS.
* Patients on IV DMT will not be included in the study.
* Non-English speaking patients

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Ann Yeh, MD, Principal Investigator — University of Toronto, The Hospital for Sick Children
Locations (13):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Loma Linda University, Loma Linda, California
  - The Regents of the University of California, San Francisco, San Francisco, California
  - University of Colorado at Denver, Denver, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Yeh EA, Chiang N, Darshan B, Nejati N, Grover SA, Schwartz CE, Slater R, Finlayson M; Pediatric MS Adherence Study Group. Adherence in Youth With Multiple Sclerosis: A Qualitative Assessment of Habit Formation, Barriers, and Facilitators. Qual Health Res. 2019 Apr;29(5):645-657. doi: 10.1177/1049732318779039. Epub 2018 Jun 17. PMID 29911511
- [Derived] Yeh EA, Grover SA, Powell VE, Alper G, Banwell BL, Edwards K, Gorman M, Graves J, Lotze TE, Mah JK, Mednick L, Ness J, Obadia M, Slater R, Waldman A, Waubant E, Schwartz CE; Pediatric MS Adherence Study Group. Correction to: Impact of an electronic monitoring device and behavioural feedback on adherence to multiple sclerosis therapies in youth: results of a randomized trial. Qual Life Res. 2018 Apr;27(4):1117. doi: 10.1007/s11136-017-1773-4. PMID 29274015
- [Derived] Yeh EA, Grover SA, Powell VE, Alper G, Banwell BL, Edwards K, Gorman M, Graves J, Lotze TE, Mah JK, Mednick L, Ness J, Obadia M, Slater R, Waldman A, Waubant E, Schwartz CE; Pediatric MS Adherence Study Group. Impact of an electronic monitoring device and behavioral feedback on adherence to multiple sclerosis therapies in youth: results of a randomized trial. Qual Life Res. 2017 Sep;26(9):2333-2349. doi: 10.1007/s11136-017-1571-z. Epub 2017 Apr 9. PMID 28393317
- [Derived] Schwartz CE, Grover SA, Powell VE, Noguera A, Mah JK, Mar S, Mednick L, Banwell BL, Alper G, Rensel M, Gorman M, Waldman A, Schreiner T, Waubant E, Yeh EA. Risk factors for non-adherence to disease-modifying therapy in pediatric multiple sclerosis. Mult Scler. 2018 Feb;24(2):175-185. doi: 10.1177/1352458517695469. Epub 2017 Feb 1. PMID 28273780

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were assigned to a study arm after completion of the enrollment visit. Thus, any participants who consented but did not complete the enrollment visit were not assigned to a study arm.
Groups:
- Behavioural Intervention/Feedback: The behavioral interventionist will contact the patient and parent by email and telephone to schedule a telephone call to review the downloaded adherence information and discuss barriers experienced by the patient/parent using a standard script. The behavioral feedback will be administered three times: at 1-, 2- and 3-months post-baseline.
  Motivational Interview
- Video Attention Control: The patients in this arm of the study will be emailed a link to an educational video about Pediatric MS and therapy for MS at three time points: 1-, 2-, and 3-months post-baseline.
  Video Attention Control
Period: Overall Study
Arm/Group | Behavioural Intervention/Feedback | Video Attention Control
Started | 31 | 32
Completed | 25 | 27
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Population: Analysis population included those participating the full trial (had two or three time points)
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioural Intervention/Feedback | Video Attention Control | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 27 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.32 (1.81) | 15.76 (2.52) | 16.03 (2.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 7 | 11 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 11 | 23
  Other | 13 | 16 | 29
Region of Enrollment [Number; unit: participants]
  Canada | 13 | 10 | 23
  United States | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Adherence in Subjects (Objective Measure)
Description: Objective measures included: (A) pharmacy refill data provided by site coordinators for 12 months prior to study entry and for 6 months post-study entry and (B) the MEMS cap, an EM device (MEMS, AARDEX) that captures each time the patient discards a needle from their injection or opens their pill bottle. Adherence information from MEMS caps is downloaded and stored on a secured web-platform (medAmigo™). These data were used to compile drug-dosing history data and to calculate medication adherence during the course of the study.
Time Frame: Baseline, 3 months, 6 months
Population: Behavioural Intervention /Feedback and Video Attention Control Arms were combined to look at changes in adherence over time (baseline, 3-months and 6-months)
Measure: Mean (Standard Deviation); unit: Proportion of doses (actual vs expected)
Arm/Group | Baseline | 3-month Follow up | 6-month Follow up
Number analyzed (Participants) | 51 | 52 | 49
Proportion of doses (actual vs expected)
  Pharmacy refill adherence | 0.95 (0.12) | 0.86 (0.20) | 0.85 (0.22)
  MEMs cap adherence: number analyzed (Participants) | 46 | 47 | 45
  MEMs cap adherence | 0.81 (0.22) | 0.82 (0.18) | 0.66 (0.32)

2. Primary Outcome: Change in Level of Adherence in Subjects (Parent- and Patient-Reported): MSTAQ
Description: Multiple Sclerosis Treatment Adherence Questionnaire (MSTAQ): Assesses missed doses, side effects and barriers of taking DMTs, and behavioral coping strategies used (e.g., icing the injection site, taking pain medication) over the past four weeks. We adapted the MSTAQ to include both oral and injectable medications. We used a standardized scoring algorithm (0-100), where higher scores reflected higher numbers of missed doses, side effects, barriers, or behavioral coping strategies. Subjects completed only the barriers items, and the parent completed all items.
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baseline | 3-month Follow up | 6-month Follow up
Number analyzed (Participants) | 47 | 45 | 47
Score on a scale
  Parent MSTAQ missed doses | 0.06 (0.18) | 0.07 (0.19) | 0.07 (0.22)
  Parent MSTAQ behavioural coping strategies: number analyzed (Participants) | 35 | 33 | 34
  Parent MSTAQ behavioural coping strategies | 49.64 (9.58) | 49.24 (8.28) | 49.33 (10.76)
  Parent MSTAQ side effects: number analyzed (Participants) | 37 | 34 | 35
  Parent MSTAQ side effects | 50.03 (9.63) | 49.48 (9.58) | 49.04 (10.63)
  Parent MSTAQ barriers: number analyzed (Participants) | 47 | 41 | 46
  Parent MSTAQ barriers | 50.12 (10.42) | 48.66 (8.60) | 49.31 (9.74)
  Patient MSTAQ barriers: number analyzed (Participants) | 45 | 41 | 46
  Patient MSTAQ barriers | 48.88 (9.22) | 50.40 (9.57) | 50.09 (10.90)

3. Secondary Outcome: Quality of Life and Psychosocial Outcomes (Parent- and Patient-Reported): PedsQL
Description: Pediatric Quality of Life Inventory (PedsQL): A 23-item tool with subscales for physical, social, emotional, and school functioning. The PedsQL has documented reliability and validity, and has been used in a large number of pediatric quality-of-life studies. Subscale scores range from 0 to 100 with higher scores representing better functioning.
Time Frame: Baseline, 3 months, 6 months
Population: The number analyzed may differ from the overall number analyzed when not all participants completed each measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baseline | 3-month Follow up | 6-month Follow up
Number analyzed (Participants) | 52 | 48 | 49
Score on a scale
  Parent: PedsQL physical functioning: number analyzed (Participants) | 51 | 48 | 49
  Parent: PedsQL physical functioning | 80.39 (22.32) | 76.69 (24.60) | 80.93 (21.34)
  Parent: PedsQL emotional functioning: number analyzed (Participants) | 51 | 48 | 49
  Parent: PedsQL emotional functioning | 73.04 (21.61) | 73.23 (19.03) | 72.30 (20.09)
  Parent: PedsQL social functioning: number analyzed (Participants) | 51 | 48 | 49
  Parent: PedsQL social functioning | 82.35 (18.56) | 84.27 (17.74) | 84.72 (20.06)
  Parent: PedsQL school functioning: number analyzed (Participants) | 51 | 48 | 49
  Parent: PedsQL school functioning | 68.24 (16.27) | 68.13 (18.24) | 68.27 (19.75)
  Patient: PedsQL physical functioning | 82.23 (17.85) | 81.51 (15.95) | 79.21 (20.64)
  Patient: PedsQL emotional functioning: number analyzed (Participants) | 52 | 47 | 49
  Patient: PedsQL emotional functioning | 71.15 (20.52) | 69.57 (21.44) | 66.63 (20.50)
  Patient: PedsQL social functioning | 83.56 (15.85) | 80.63 (19.34) | 82.65 (20.36)

4. Other Pre Specified Outcome: Well-Being
Description: Autonomy and Environmental Mastery subscale scores (Ryff Scales of Psychological Well-Being) will be compared at baseline, three months, and six months between the two study arms.
Time Frame: baseline, three months, and six months
Reporting Status: Not Posted

5. Primary Outcome: Change in Level of Adherence in Subjects (Parent- and Patient-Reported): Morisky
Description: Morisky Adherence Scale (Morisky): A widely used 8-item patient-/parent-reported measure with documented reliability and validity. Total scores range from 0 to 8.The following scoring algorithm was used: 8 = high adherence, 6-7 = medium adherence, and <6=low adherence.
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baseline | 3-month Follow up | 6-month Follow up
Number analyzed (Participants) | 52 | 48 | 49
Score on a scale
  Parent Morisky: number analyzed (Participants) | 49 | 47 | 49
  Parent Morisky | 6.28 (1.46) | 6.40 (1.50) | 6.20 (1.85)
  Patient Morisky | 5.93 (1.74) | 6.00 (1.82) | 5.94 (1.91)

6. Primary Outcome: Change in Level of Adherence in Subjects (Parent- and Patient-Reported): Parental Involvement
Description: Parental involvement in DMT administration (Parental Involvement): Percentage of time the parent reported (1) reminding the child to take her/his DMT; (2) being present when the child took her/his DMT; and (3) administering the child's DMT.
Time Frame: Baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Baseline | 3-month Follow up | 6-month Follow up
Number analyzed (Participants) | 51 | 48 | 49
Percentage of time
  Parent remind | 44.61 (38.83) | 37.50 (37.90) | 33.16 (34.76)
  Parent present | 65.20 (37.11) | 55.21 (39.26) | 57.14 (39.53)
  Parent administer | 36.27 (41.33) | 32.81 (41.95) | 30.10 (40.82)

7. Secondary Outcome: Quality of Life and Psychosocial Outcomes (Parent- and Patient-Reported): MSNQ
Description: Multiple Sclerosis Neuropsychological Screening Assessment Questionnaire (MSNQ): Neurocognitive Functioning will be assessed using the informant-report version of the Multiple Sclerosis Neuropsychological Screening Assessment Questionnaire (MSNQ). This 15-item tool has documented high test-retest stability, predictive validity, and construct validity. Informant reports are documented to be reliably correlated with cognitive dysfunction and be less biased by patient depression. Total scores range from 0 to 60 with a higher score indicating worse cognitive functioning.
Time Frame: Baseline, 3 months, 6 months
Population: The number analyzed may differ from the overall number analyzed when not all participants completed each measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Baseline | 3-month Follow up | 6-month Follow up
Number analyzed (Participants) | 49 | 47 | 49
Score on a scale | 17.90 (13.42) | 17.55 (12.41) | 20.24 (14.60)

ADVERSE EVENTS:
Arm/Group | Behavioural Intervention/Feedback | Video Attention Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No